CLINICAL TRIAL: NCT00305643
Title: A Multicenter Phase III Placebo-Controlled Trial of Celecoxib for Prevention of Capecitabine-Induced Palmar/Plantar (Hand/Foot) Syndrome in Patients With Metastatic Breast and Colorectal Cancer
Brief Title: Celecoxib in Preventing Hand/Foot Syndrome Caused By Capecitabine With Metastatic Breast or Colorectal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to low accrual. No data analyzed.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2005-0328; MDA-CCC-0326 (Other: NCI); MDA-2005-0328 (Other: NCI); CDR0000458042 (Registry Identifier: NCI)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer; Colorectal Cancer; Pain
Keywords: Hand-Foot Syndrome; cancer-related problem/condition; drug/agent toxicity by tissue/organ; pain; palmar-plantar erythrodysesthesia; stage IV breast cancer; male breast cancer; recurrent breast cancer; stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; Celecoxib; Celebrex; Capecitabine; Xeloda
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Pain; Hand-Foot Syndrome; Drug-Related Side Effects and Adverse Reactions; Breast Neoplasms, Male; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Celecoxib; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Celecoxib + Capecitabine (Experimental): Celecoxib 200 mg given orally twice/day along with standard capecitabine treatment (Initial dose of 750-1500 mg/m^2 orally twice/day).
  Interventions: Drug: Capecitabine; Drug: Celecoxib; Procedure: Radiation Therapy
- Arm II: Placebo + Capecitabine (Placebo Comparator): Placebo with standard capecitabine treatment (Initial dose of 750-1500 mg/m^2 orally twice/day)
  Interventions: Drug: Capecitabine; Procedure: Radiation Therapy; Drug: Placebo

INTERVENTIONS:
Drug: Capecitabine — Initial dose of 750-1500 mg/m^2 orally twice a day for each 21 day cycle.
  Other Names: Xeloda
Drug: Celecoxib — 200 mg given orally twice a day for each 21 day cycle.
  Other Names: Celebrex
  Arms: Arm I: Celecoxib + Capecitabine
Procedure: Radiation Therapy — Some patients may undergo radiation therapy 5 days a week for 5-6 weeks, and receive oral capecitabine twice daily 5 days a week. Following completion of radiotherapy, patients may continue oral capecitabine once daily on days 1-14.
  Other Names: RT; XRT
Drug: Placebo — Oral placebo twice daily on days 1-21
  Arms: Arm II: Placebo + Capecitabine

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with capecitabine may kill more tumor cells. Celecoxib may prevent or lessen hand-foot syndrome caused by capecitabine.

PURPOSE: This randomized phase III trial is studying how well celecoxib works in preventing hand/foot syndrome caused by capecitabine in patients with metastatic breast or colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of celecoxib in reducing the incidence and severity of hand/foot syndrome caused by capecitabine in patients with metastatic breast cancer or colorectal cancer.

OUTLINE: This is a placebo-controlled, randomized, double-blind, multicenter study. Patients are stratified according to metastatic disease (breast vs colorectal), ECOG performance status (0 or 1 vs 2), prior chemotherapy (yes vs no).

Patients receive 1 of 2 treatment regimens.

* Regimen A (concurrent radiotherapy): Patients undergo radiotherapy 5 days a week for 5-6 weeks and receive oral capecitabine twice daily 5 days a week. Following completion of radiotherapy, patients may continue oral capecitabine as in regimen B.
* Regimen B (no radiotherapy): Patients receive oral capecitabine once daily on days 1-14. Courses repeat every 21 days.

Patients are also randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral celecoxib twice daily on days 1-21.
* Arm II: Patients receive oral placebo twice daily on days 1-21. In both arms, treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 342 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic colorectal cancer or breast cancer who are scheduled*** to receive capecitabine with an initial dose in the range of 750-1500 mg/m2** twice daily (total daily dose in the range of 1500-3000 mg/m2) alone or in combination with one or more other agents. ***Patients may enter the study after having received capecitabine for up to 21 days prior to study entry. **Doses may be rounded upward or downward per physician discretion to utilize 500mg tablets.
2. Patients with either metastatic colorectal or metastatic breast cancer may have received any number or type of prior treatment regimens for metastatic disease or they may have received no prior treatment for metastatic disease.
3. Men and women from all ethnic and racial groups.
4. >/= 18 years old
5. Eastern Cooperative Oncology Group (ECOG) Performance Status </= 2
6. Adequate organ function: a. Total bilirubin </= 1.5 * the institutional upper-normal limits (IUNL) b. aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) </= 2.5 * IUNL c. Patients with liver mets AST/(SGOT) and/or ALT(SGPT) < 5 * IUNL d. Alkaline phosphatase </= 5 * IUNL e. Creatinine Clearance > 50 ml/min
7. Adequate bone marrow function: (a) Leukocytes >/= 3,000/microL; (b) Absolute neutrophil count >/= 1,500/microL; (c) Platelets >/= 100,000/microL
8. Women of childbearing age and all men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.
9. Negative pregnancy test for women of childbearing age.
10. Must have the ability to understand and the willingness to provide a written informed consent to participate in the study.
11. Controlled brain metastasis (i.e. stereotactic surgery, surgery steroids, anticonvulsants).

Exclusion Criteria:

1. History of allergies to sulfonamide, aspirin, any NSAID (Nonsteroidal anti-inflammatory drugs)or 5FU or any COX-2 inhibitor.
2. Any regular use of COX-2 inhibitors, NSAIDS or aspirin >325 mg more than twice a week.
3. Pregnancy or lactation.
4. History of significant neurological or psychiatric disorders that would impede giving consent, treatment or follow-up.
5. Any serious illness or medical condition: uncontrolled congestive heart failure, uncontrolled hypertension or arrhythmia, active angina pectoris, any history of myocardial infarction, stroke or transient ischemic attack (TIA).
6. Serious uncontrolled active infection.
7. Patients who cannot comply with taking and documenting oral study medications.
8. History of active peptic ulcer disease or upper gastrointestinal (GI) bleed within 12 months of enrollment.
9. Use of warfarin.
10. Patients with uncontrolled brain metastasis.
11. Patients may have had prior Hand-foot syndrome (HFS) but it must be completely resolved for >/= 4 weeks.
12. No concurrent radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kopetz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (14):
- United States (13):
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - Hematology Oncology Associates of Central New York, PC - Northeast Center, East Syracuse, New York
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - CCOP - Greenville, Greenville, South Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Scott and White Cancer Institute, Temple, Texas
  - CCOP - Northwest, Tacoma, Washington
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- MBCCOP - San Juan, San Juan, Puerto Rico

REFERENCES:
- See also: Clinical trial summary, the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 27, 2006 to October 06, 2008 from various medical clinics and institutions representing the Community Clinical Oncology Program (CCOP).
Pre-assignment Details: Study terminated due to slow accrual.
Groups:
- Arm I: Celecoxib + Capecitabine: Arm I: Celecoxib 200 mg given orally twice/day along with standard capecitabine treatment (Initial dose of 750-1500 mg/m^2 orally twice/day).
- Arm II: Placebo + Capecitabine: Arm II: Placebo with standard Capecitabine treatment (Initial dose of 750-1500 mg/m^2 orally twice/day).
Period: Overall Study
Arm/Group | Arm I: Celecoxib + Capecitabine | Arm II: Placebo + Capecitabine
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Celecoxib + Capecitabine | Arm II: Placebo + Capecitabine | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Full Range); unit: years] | 61 [47 to 76] | 66 [50 to 83] | 63 [47 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
  Puerto Rico | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hand/Foot Syndrome (HFS) > Grade 1 at 16 Weeks Based on the CTC 3.0 Criteria.
Description: The primary classification of palmar planter erythrodysethesia according to National Cancer Institute Common Toxicity Criteria (CTC) 3.0 criteria used to determine the incidences of > grade 1 hand and foot syndrome (HFS) by 16 weeks from the commencement of therapy.
Time Frame: At 16 Weeks, with evaluations and blood test every 3 weeks.
Population: No analysis could be performed due to low accrual and no participants reaching the 16 week mark.
Arm/Group | Arm I: Celecoxib + Capecitabine | Arm II: Placebo + Capecitabine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Hand/Foot Syndrome (HFS) > Grade 1 at 16 Weeks Based on WHO Criteria.
Description: A secondary classification of palmar planter erythrodysethesia according to World Health Organization (WHO) criteria will be used for determination of the incidences of > grade 1 HFS by 16 weeks from the commencement of therapy.
Time Frame: At 16 Weeks
Population: No analysis could be performed due to low accrual and no participants reaching the 16 week mark.
Arm/Group | Arm I: Celecoxib + Capecitabine | Arm II: Placebo + Capecitabine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection from baseline to 30 days following discontinuation of study drug. Overall study period: 2 years and 6 months
Arm/Group | Arm I: Celecoxib + Capecitabine | Arm II: Placebo + Capecitabine
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Celecoxib + Capecitabine (N=6) | Arm II: Placebo + Capecitabine (N=5)
Cardiac Ischemia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Celecoxib + Capecitabine (N=6) | Arm II: Placebo + Capecitabine (N=5)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 1 (1)
Hand-foot (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mucositis (clinical exam) - Oral cavity
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lab - Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lumbar Spine Range of Mobility Decrease (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neuropathy - Motor (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy - Sensory (Nervous system disorders) | 0 (0) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - Limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Renal - Other (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain - Other (General disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to low accrual in this trial, no outcome measures were evaluable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No